CLINICAL TRIAL: NCT03956875
Title: Yoga for Aromatase Inhibitor-related Knee Pain Relief in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CMUH107-REC3-102
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Breast Cancer; Aromatase Inhibitor; Yoga; Knee Pain
MeSH Terms: conditions — Breast Neoplasms | interventions — Yoga; Massage

STUDY DESIGN:
Intervention Model Description: The investigators designed a crossover study, a total of 60 patients divided equally to control group (massage for 6 weeks in home care) and treatment group (Yoga treatment for 12 times/6 weeks).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- yoga (Active Comparator): Yoga treatment
  Interventions: Other: yoga
- massage (Placebo Comparator): massage
  Interventions: Other: yoga

INTERVENTIONS:
Other: yoga — yoga is a mind-body practice that guides the body through a series of poses and breathing exercises
  Other Names: massage

SUMMARY:
The purpose of the study was to investigate the therapeutic effect of Yoga on aromatic inhibitor-induced chronic knee pain in patients with breast cancer.

DETAILED DESCRIPTION:
Estrogen plays a critical role in breast cancer growth in pre-and post-menopausal women. The aromatic catalyzer has relationship with biosynthesis of estrogen, therefore, aromatic inhibitors became as a standard therapy of breast cancer in post-menopausal women. Arthralgia and joint stiffness are most common side effect in aromatic inhibitor treatment. Yoga is benefit for the patients with chronic pain improvement, and also can improve quality of life. Therefore, the purpose of the present study was to investigate the therapeutic effect of Yoga on aromatic inhibitor-induced chronic knee pain in patients with breast cancer.The investigators designed a crossover study, a total of 60 patients divided equally to control group (massage for 6 weeks in home care) and treatment group (Yoga treatment for 12 times/6 weeks). There is two weeks wash out period after finishing 6 weeks treatment, and then the patients in control group changed to treatment, in contrast, the patients in the treatment changed to control group. The assessment time was pre-treatment (vision 1), finishing 6 weeks treatment (vision), finishing 6 weeks treatment after crossover (vision 3). The major assessment was brief pain inventory scores changed The results in the present study predict Yoga treatment for 6 weeks can improve aromatic inhibitor-induced knee pain and also can improve quality of life in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with breast cancer and is taking an aromatic ring enzyme inhibitor. Knee joint pain for more than three months. Ages are over 20 years old and under 70 years old.

Exclusion Criteria:

At the same time, there are multiple sources of pain associated with non-breast cancer, such as visceral pain, traumatic pain, which must be excluded by the moderator.

Addicted drug abusers, subject to the judgment of the host. Women who may be pregnant, pregnant women, within three months after childbirth.

Have a serious mental illness or an unstable mental state, which will affect the clinical assessment.

Severe hearing impairment, visual impairment, or dementia. It is not easy to measure by the host.

Limb edema and severe skin damage are not suitable for yoga practitioners by the physician.

The spinal lesions are excessively severe, affecting the normal function of the operation, and the test cannot be completed.

Have been a yoga practitioner for nearly a month, or a regular exerciser for over 90 minutes per week for the past month.

Cancer has been transferred (stage IV)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
womac questionnaire | 3 minutes
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis.

SECONDARY OUTCOMES:
M.E.A.D (Meridian Energy Analysis Device) | 5minutes
  The instrument mainly detects 24 representative points of the twelve meridians around the human body. The bioelectrical resistance of each meridian is measured by the test rod to evaluate the conductivity of each meridian, and the physiology of the subject is analyzed by computer. situation.

CONTACTS AND LOCATIONS:
Locations (1):
- Ching-Liang Hsieh, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
undecided